CLINICAL TRIAL: NCT02177981
Title: A Randomized, Double-Blind, Controlled Clinical Trial: Impact of Remote Ischemic Preconditioning Preceding Coronary Artery Bypass Grafting on Inducing Neuroprotection
Brief Title: Impact of Remote Ischemic Preconditioning Preceding Coronary Artery Bypass Grafting on Inducing nEuroprotection
Acronym: RIPCAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zagreb (Other)
Collaborators: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Hrvoje Gasparovic, MD, PhD, Associate professor, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 57./3./1.
Record Dates: First submitted 2014-04-07; First posted 2014-06-30 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Brain Ischemia; Postoperative Confusion
Keywords: Remote Ischemic Preconditioning; Coronary Artery Bypass Grafting; Diffusion Weighted Magnetic Resonance Imaging; Resting State Functional Magnetic Resonance Imaging; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Brain Ischemia; Postoperative Cognitive Complications

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote ischemic preconditioning (Active Comparator): A blood pressure cuff will be placed on the left arm and three cycles of 5 min ischemia followed by 5 min reperfusion will be applied.
  Interventions: Procedure: Remote ischemic preconditioning
- Control (Sham Comparator): The cuff will be placed around the arm but not inflated.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — A blood pressure cuff will be placed on the left arm and three cycles of 5 min ischemia followed by 5 min reperfusion will be applied.
  Arms: Remote ischemic preconditioning
Procedure: Control — The cuff will be placed around the arm but not inflated.
  Arms: Control

SUMMARY:
Coronary artery disease (CAD) is the leading cause of death worldwide. Patients with severe CAD are often treated with coronary artery bypass grafting (CABG). Novel treatment strategies need to be pursued to respond to the continuous increase in the risk profile of contemporary CABG patients. Surgical myocardial revascularization is commonly performed with the use of cardiopulmonary bypass (CPB). Neurological impairment following CABG may take on the form of a new-onset motor deficit or postoperative cognitive dysfunction. The former is rare, but potentially devastating. Conversely, declines in attention, memory and fine motor skills can frequently be documented.

Ischemic preconditioning is a phenomenon of an endogenous protective response to organ ischemia, which is triggered by brief cycles of nonlethal ischemia and reperfusion in tissues known to be more resistant to ischemic insults. In clinical practice remote ischemic preconditioning (RIPC) is achieved by inflicting short periods of ischemia with intermittent restitution of flow to the upper extremity. This intervention has been shown to be effective in the reduction of myocardial injury in cardiac surgical patients. The hypothesis tested in this research proposal is that RIPC will decrease the extent of postoperative neurological injury following CABG.

In this research project, 70 patients scheduled for an elective CABG will be recruited at a single center. They will be randomly allocated to either undergo RIPC (intervention arm) or a sham procedure (control arm). Inflating a blood pressure cuff to 200 mmHg for 5 min will induce RIPC, thereby inducing a brief period of ischemia. This will be followed by a 5-minute arm reperfusion. In total, three cycles of arm ischemia and reperfusion will be induced in this fashion.

All patients will undergo pre- and post-procedural magnetic resonance imaging (MRI) of the brain, as well as neurocognitive testing. The array of MRI tools that will be used for the quantification of brain injury will include fluid attenuated inversion recovery, diffusion weighted and susceptibility weighted imaging, coupled with resting state functional MRI.

The investigators aim to determine whether RIPC can reduce the adverse impact of CPB on neurological outcome as evaluated by MRI detectable brain ischemia and neurocognition.

DETAILED DESCRIPTION:
Coronary artery bypass grafting (CABG) is very effective in the management of complex coronary artery disease (CAD). Cardiopulmonary bypass (CPB) is commonly employed to achieve a still and bloodless field, which facilitates the creation of technically impeccable coronary anastomoses. Multiple adverse effects that stem from exposure of blood to a non-endothelial surface contrast the clear benefit of CPB. Neurological damage remains one of the most dreaded complications following CABG. While the incidence of new focal motor deficits is low, postoperative neurocognitive dysfunction (POCD) is seen commonly. The increasing risk profile of contemporary CABG patients makes neuroprotective strategies progressively more important.

Ischemic preconditioning is an endogenous protective response triggered by brief episodes of nonlethal ischemia and reperfusion. In clinical practice remote ischemic preconditioning (RIPC) is achieved by inducing short periods of ischemia of the upper extremity, followed by restitution of flow. This non-pharmacological strategy for inducing ischemic tolerance is cost-free and non-invasive, with potentially wide clinical applicability.

The "Impact of Remote Ischemic Preconditioning preceding Coronary Artery bypass Grafting on inducing nEuroprotection (RIPCAGE) trial" will recruit 70 patients scheduled for elective CABG at a single academic center. The hypothesis tested in this research proposal is that RIPC will decrease the extent of postoperative neuronal damage and lead to a reduction in POCD among CABG patients. Specifically, the investigators aim to determine whether RIPC can reduce magnetic resonance imaging (MRI) detectable brain damage and attenuate the neurocognitive decline universally seen in patients after CABG.

The primary composite outcome will consist of a composite of new ischemic lesions on brain MRI and POCD.

The secondary endpoints will be the following:

1. Brain connectivity profiles on resting-state functional MRI (rs-fMRI).
2. Pooled ischemic volumes of new diffusion-weighted imaging (DWI) hyperintensity.
3. Percent declines of components in individual neurocognitive tests.

Patients will be randomly allocated in a 1:1 ratio to either receive RIPC or no intervention (control group). In the intervention arm, transient upper extremity ischemia will be induced after induction of anesthesia by inflating a blood pressure cuff to 200 mmHg for 5 min, followed by a 5 min cuff deflation. This sequence will be repeated 3 times. Patients in the control group will also have a blood pressure cuff placed, but it will not be inflated. All patients will undergo preoperative neurocognitive testing coupled with baseline brain MRI. The neurocognitive evaluation will consist of the Montreal Cognitive Assessment (MoCA) test and the Trail Making Test (TMT). Decreased cognitive function for each test will be defined as an individual decrease of at least 1 standard deviation of the group baseline mean for that test. POCD will be defined as a decrease in two or more tests. The patients will have a repeat neurocognitive evaluation prior to discharge from hospital.

Standard MRI sequences will be performed in all patients. DWI will be utilized for volumetric analysis of brain tissue exhibiting stigmata of ischemic injury. The timing of apparent diffusion coefficient quantification will be standardized to postoperative day 7, as it normalizes over time. Additional MRI sequences will include susceptibility weighted imaging (SWI) and diffusion tensor imaging (DTI). Resting state functional MRI will be performed in order to investigate the coordination of activity across brain networks. Pre- and postprocedural rs-fMRI data will be subsequently compared with each other. Disruption in the connectivity of neural circuits induced by the operation will be thereby be objectivized.

Patients will be followed for a total of 3 months, during which time all adverse events will be recorded and adjudicated by an independent clinical events committee.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with multi-vessel coronary artery disease undergoing primary, elective on-pump CABG
* Written informed consent

Exclusion Criteria:

* Prior stroke, transient ischemic attack or reversible ischemic neurologic deficit
* Stenosis of the internal carotid artery (>50%)
* Significant peripheral arterial disease affecting the upper limbs
* Acute coronary syndrome within 30 days prior to surgery
* Inability to provide consent
* Postoperative exclusion criteria will be limited to contraindications to follow-up MRI (such as pacemaker dependence)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Composite structural and functional neurological outcome | 7 days
  New ischemic lesions on brain MRI and postoperative neurocognitive dysfunction

SECONDARY OUTCOMES:
Brain connectivity profiles | 7 days
  Changes between pre- and postoperative resting state functional MRI expressed as continuous variables and subsequently compared among the intervention and control arms
Peri-operative brain injury | 7 days
  Volumetric quantification of areas of new diffusion-weighted imaging hyperintensity in individual patients
Postoperative neurocognitive decline | 7 days
  Percent declines in individual neurocognitive tests

CONTACTS AND LOCATIONS:
Overall Officials: Hrvoje Gašparović, MD, PhD, Study Chair — University of Zagreb School of Medicine
Locations (1):
- University Hospital Centre Zagreb, Zagreb, City of Zagreb, Croatia

REFERENCES:
- [Derived] Gasparovic H, Kopjar T, Rados M, Anticevic A, Rados M, Malojcic B, Ivancan V, Fabijanic T, Cikes M, Milicic D, Gasparovic V, Biocina B. Impact of remote ischemic preconditioning preceding coronary artery bypass grafting on inducing neuroprotection (RIPCAGE): study protocol for a randomized controlled trial. Trials. 2014 Oct 27;15:414. doi: 10.1186/1745-6215-15-414. PMID 25348157